CLINICAL TRIAL: NCT04834830
Title: Evaluation and Importance of the PD-1/PD-L1 and the IL-10/IL-10R Axis in Malignant and Benign Pleural Effusions - a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Daniela Gompelmann, Prof. Dr. med., University of Vienna
Other Study IDs: Version 1.1 26.01.2021
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pleural effusion: In patients with pleural effusion and indication for diagnostic and/or therapeutic procedures (thoracocentesis, drainage of fluid, indwelling pleural catheter (IPC) management, and/or video-assisted thoracoscopic surgery), pleural fluid will be examined for various cytokines and PD1-lymphoctyes.
  Interventions: Diagnostic Test: Pleural effusion will be examined for various cytokines and PD1-lymphocytes.

INTERVENTIONS:
Diagnostic Test: Pleural effusion will be examined for various cytokines and PD1-lymphocytes. — Examination of pleural effusion

SUMMARY:
The aim of this study is to evaluate the concentrations of interleukin-2, interleukin-10, interferon-gamma, PD1+ lymphocytes, and the interleukin-10 receptor expression in malignant and benign effusions.

DETAILED DESCRIPTION:
In this prospective trial, 80 patients with pleural effusions and indication for thoracocentesis, drainage, indwelling pleural catheter (IPC) management and/or video-assisted thoracoscopic surgery are enrolled. The pleural effusion will be examined for different cytokines, cytokine-receptors, PD1-lymphocytes and CD4+/CD25+/Foxp3+ regulatory T cell.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* radiologically confirmed pleural effusion with an indication for puncture, pleural drain insertion, or video-assisted thoracoscopy for diagnostic and/or therapeutic reasons
* Signed declaration of consent

Exclusion Criteria:

* Withdrawal or cessation of participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with malignant or benign pleural effusions requiring diagnostic and/or therapeutic procedures including thoracocentesis, drainage insertion, indwelling pleural catheter (IPC) management, and/or video-assisted thoracoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
To assess and compare the concentration of various cytokines and PD1-lymphoytes in malignant and benign pleural effusions | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided